CLINICAL TRIAL: NCT06333899
Title: A Pilot Study of Lorlatinib for Treatment of Children With Newly Diagnosed High-Grade Glioma With ROS-1 (ROS Proto-Oncogene 1, Receptor Tyrosine Kinase) or ALK (Anaplastic Lymphoma Kinase) Fusion
Brief Title: Lorlatinib for Newly-Diagnosed High-Grade Glioma With ROS or ALK Fusion
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT TarGeT-L; R01FD008167 (FDA)
Record Dates: First submitted 2024-03-14; First posted 2024-03-27 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-05

CONDITIONS: High Grade Glioma; Diffuse Intrinsic Pontine Glioma; Anaplastic Astrocytoma; Infant Type Hemispheric Glioma; Glioblastoma; Glioblastoma Multiforme; WHO Grade III Glioma; WHO Grade IV Glioma; Diffuse Midline Glioma, H3K27-altered
Keywords: ALK fusion; ROS fusion; High Grade Glioma; Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Glioma; Diffuse Intrinsic Pontine Glioma; Astrocytoma; Glioblastoma | interventions — lorlatinib

STUDY DESIGN:
Intervention Model Description: Feasibility
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Lorlatinib Monotherapy (Experimental): Lorlatinib administered as monotherapy by PO (per os) or NG (nasogastric) for two 28-day cycles at 115 mg/m2/day (or maximum 200mg/dose), after which disease evaluation by Magnetic Resonance Imaging (MRI) imaging will be performed.
  Interventions: Drug: Lorlatinib
- Lorlatinib Combination with BABY POG chemotherapy (Experimental): Lorlatinib monotherapy x2 cycles followed by maintenance therapy with lorlatinib (115 mg/m2/day) and BABY-POG chemotherapy backbone (vincristine, cyclophosphamide, cisplatin) The BABYPOG chemotherapy backbone regimen will consist of six 12-week courses. Each course will consist of cycles A, A2 and B, which will be administered consecutively, in 28-day cycles for a total of 72 weeks
  Interventions: Drug: Lorlatinib; Drug: Lorlatinib with chemotherapy1
- Lorlatinib Combination with HIT-SKK chemotherapy (Experimental): Lorlatinib monotherapy x2 cycles followed by maintenance therapy with lorlatinib (115 mg/m2/day) and HIT-SKK chemotherapy backbone (cyclophosphamide, vincristine, methotrexate, carboplatin, etposide) The recommended HIT-SKK chemotherapy backbone regimen consists of modular chemotherapy cycles, three courses of 4 blocks each (Element IIS, Element IIIS/1, Element IIIS/2, and Element IVS). Each element will be administered consecutively at 2-3-week intervals. Elements IIS and IVS cycles will be repeated twice thereafter. The entire length of treatment for HIT-SKK will be approximately 42 weeks.
  Interventions: Drug: Lorlatinib; Drug: Lorlatinib with chemotherapy 2
- Lorlatinib Maintenance Therapy post RT (Experimental): Lorlatinib monotherapy x2 cycles followed by Radiation Therapy and continue lorlatnib maintenance monotherapy (115 mg/m2/day) 28 days post completion of RT for 12 cycles
  Interventions: Drug: Lorlatinib; Drug: Lorlatinib post Radiation

INTERVENTIONS:
Drug: Lorlatinib — Continue maintenance monotherapy for total 12 cycles
  Other Names: LOBRENA
Drug: Lorlatinib with chemotherapy1 — Continue lorlatinib with BABY-POG chemotherapy backbone for 72 weeks
  Other Names: LOBRENA
  Arms: Lorlatinib Combination with BABY POG chemotherapy
Drug: Lorlatinib with chemotherapy 2 — Continue lorlatinib with HIT-SKK chemotherapy backbone for 42 weeks
  Other Names: LOBRENA
  Arms: Lorlatinib Combination with HIT-SKK chemotherapy
Drug: Lorlatinib post Radiation — Continue lorlatinib monotherapy 28 days post completion of radiation therapy for 12 cycles
  Other Names: LOBRENA
  Arms: Lorlatinib Maintenance Therapy post RT

SUMMARY:
The goal of this study is to determine the response of the study drug loratinib in treating children who are newly diagnosed high-grade glioma with a fusion in ALK or ROS1. It will also evaluate the safety of lorlatinib when given with chemotherapy or after radiation therapy.

DETAILED DESCRIPTION:
This is a multi-institutional clinical trial of lorlatinib in children newly diagnosed with High Grade Glioma (HGG) harboring ROS1 (ROS Proto-Oncogene 1, Receptor Tyrosine Kinase) or ALK (anaplastic lymphoma kinase) fusions. In this pilot study, investigators will assess the disease control rate (Continued Complete Response (CCR), Complete Response (CR), Partial Response (PR), and Stable Disease (SD)) of lorlatinib, and feasibility and safety of lorlatinib administration in combination with standard chemotherapy in children with newly diagnosed HGG with ROS or ALK fusions who receive 2 cycles of lorlatinib administered orally, once daily, at 115 mg/m2/day (or maximum of 200mg/dose) for pediatric patients, and 150mg/dose for patients >18 years, continuously. Secondary objectives include overall survival (OS) and progression free survival (PFS) lorlatinib as a single agent and in combination with standard chemotherapy used in children ≤ 48 months with HGG, or post focal radiotherapy in children > 48 months of age. Children with HGG who have a CCR or CR after 2 cycles of therapy will continue to receive single agent lorlatinib for a total of 12xs 28-day cycles. Continuation of treatment beyond 12 cycles, and up to maximum 26 cycles, may be considered for patients on lorlatinib monotherapy if they are receiving clinical benefit from the study, at the discretion of the treating physician after discussion with Study Chairs. Patients with PR or SD after 2 cycles of lorlatinib monotherapy will go on to receive lorlatinib either in combination with standard backbone chemotherapy (BABYPOG or HIT-SKK, investigator's choice) or post standard radiotherapy, based on the patient's age. Patients with PD after 2 cycles will be taken off protocol therapy.

This study will be a part of the TarGeT, molecularly-guided umbrealla trial in children, adolescents, and young adults newly diagnosed with HGG, including diffuse intrinsic pontine glioma (DIPG)/diffuse midline glioma (DMG). Patients will undergo (1) upfront comprehensive tumor molecular profiling using multi-omic approach with rapid return of results, (2) stratification to biologically-targeted treatment arms to assess treatment efficacy, and (3) longitudinal evaluation of peripheral blood, cerebrospinal fluid (CSF), and/or tumor tissue as well as neuro-imaging to identify biomarkers predictive of response, recurrence, and resistance.

Based on recent trials conducted in this patient population, investigators conservatively estimate that 1 child with newly diagnosed DIPG or HGG with either ROS1 or ALK fusion will be enrolled every 2 months on this study. Patients ≤18 years will start at the recommended phase 2 dose of 115 mg/m2/day and patients >18 years will start at 150mg/dose. All patients will be treated continuously for 28 days, and one dose de-de-escalations will be allowed. A maximum of 15 eligible patients will be enrolled, anticipated over 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 12 months and ≤ 21 years of age at the time of study enrollment on TarGeT-SCR.
2. Diagnosis:

   Patients with newly diagnosed high-grade glioma (HGG), including diffuse intrinsic pontine gliomas (DIPG), whose tumors harbor an ALK or ROS-1 fusion alteration are eligible. Patients must have had histologically verified high-grade glioma from diagnostic biopsy or resection. For the diagnosis of DIPG, patients must have a tumor with pontine epicenter and diffuse involvement of at least 2/3 of the pons, with histopathology consistent with diffuse WHO Grade 2-4. All other HGGs must be Grade 3 or 4.
3. Disease Status:

   Patients with disseminated DIPG or HGG are eligible only if the patient is to receive chemotherapy only, i.e. no craniospinal RT is intended to be given. MRI of spine must be performed if disseminated disease is suspected clinically by the treating physicians. Patients with primary spinal tumors are eligible only if the patient is to receive either chemotherapy or focal radiation therapy, i.e., no craniospinal RT is intended to be given. Patients with leptomeningeal disease only, with no definitive identifiable primary tumor, and documented ALK or ROS-1 fusion, must be discussed with the Study Chair on a case-by-case basis.
4. Performance Level:

   Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age (See Appendix I). Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
5. Prior Therapy:

   * Patients must not have received any prior anti-cancer chemotherapy.
   * Prior use of corticosteroids is allowed (see below Exclusion Criteria)
6. Organ Function Requirements 6.1 Adequate Bone Marrow Function Defined as:

   * Peripheral absolute neutrophil count (ANC) ≥ 1000/μL
   * Platelet count ≥ 100,000/μL (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
   * Hemoglobin >8 g/dL (may receive transfusions) 6.2 Adequate Renal Function Defined as:
   * Serum creatinine within normal institutional limits OR Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 6.3 Adequate Liver Function Defined as:
   * Total bilirubin ≤ 2 × institutional upper limit of normal
   * AST(aspartate aminotransferase)/ALT(alanine transaminase) ≤ 2.5 × institutional upper limit of normal 6.4 Adequate Pulmonary Function Defined as: Pulse oximetry > 94% on room air if there is clinical indication for determination (e.g. dyspnea at rest).

6.5Adequate Cardiac Function Defined as: QTc ≤ 470 msec (by Bazett formula) 6.6 Adequate Neurologic Function Defined as: Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled.

6.7 Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

1. Pregnant or breast-feeding women will not be entered on this study due to unknown risks of fetal and teratogenic adverse events as seen in animal/human studies. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

   Females of reproductive potential must use an effective non-hormonal method of contraception, since lorlatinib can render hormonal contraceptives ineffective, during study treatment and for at least 6 months after the final dose. Males with female partners of reproductive potential must use effective contraception during treatment with lorlatinib and for 3 months after the final dose.
2. Concomitant Medications

   * Investigational Agents/Drugs: Patients who have previously received or are currently receiving another investigational drug are not eligible.
   * Anti-cancer Agents: Patients who have previously received or are currently receiving other anti-cancer agents, including chemotherapy, immunotherapy, monoclonal antibodies, biologic or targeted therapy, are not eligible
3. Infection: Patients must not have any active, uncontrolled systemic bacterial, viral or fungal infection.
4. Patients who have received prior solid organ transplantation are not eligible.
5. Patients must not have malabsorption syndrome or other condition affecting oral absorption.
6. Patients must not be receiving any treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor or inducer. Discontinue strong CYP3A inducers for 3 plasma half-lives of the strong CYP3A inducer prior to treatment with loraltinib. Moderate inducers of CYP3A4 should be avoided
7. Avoid concomitant use of lorlatinib with certain CYP3A substrates, for which minimal concentration changes may lead to serious therapeutic failures. If concomitant use is unavoidable, increase the CYP3A substrate dosage in accordance with approved product labeling.
8. P-glycoprotein (P-gp) substrates: Lorlatinib is considered a moderate P-gp inducer. Co-administration of lorlatinib with P-gp substrates including but not limited to digoxin should be avoided as the concentration of these drugs may be reduced by lorlatinib.
9. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.
10. Patients with a known personal history of acute or chronic severe psychiatric disorders or current history of suicidal ideation and history of suicide attempt.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-03 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2035-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | Day 1 of treatment until the end of cycle 2 (each cycle is 28 days)
  To assess the disease control rate (Complete Response [CR], Continued Complete Response [CCR], Partial Response [PR] and Stable Disease [SD]) of lorlatinib in young children with newly diagnosed high-grade glioma with ALK or ROS1 fusion after 2 cycles of lorlatinib monotherapy.
Number of participants with lorlatinib-related adverse events as assessed by CTCAE v5.0 | From Day 1 of protocol treatment through 30 days following end of protocol treatment
  Assess and further characterize the safety and toxicity of lorlatinib in pediatric patients newly diagnosed with HGG with a fusion in ALK or ROS. This will be achieved by calculating the number of participants with, as well as frequency and severity of, lorlatinib-related Adverse Events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) in HGG | From Day 1 of protocol treatment through 30 days following end of protocol treatment
  To assess the objective response rate (ORR) (Complete Response [CR] and Partial Response [PR]) of lorlatinib in children with newly diagnosed high-grade glioma with ALK or ROS1 fusion after 2 cycles of lorlatinib monotherapy.
Overall Survival (OS) in HGG | Day 1 of treatment until date of death due to any cause or date of last follow-up, assessed up to 60 months
  To assess overall (OS) of children with high-grade gliomas treated with a lorlatinib-containing regimen at 1, 3 and 5 years and compare it to historical data from BABYPOG and HIT-SKK.
Progression-Free Survival in HGG | Day 1 of treatment until date of Progressive Disease or death due to any cause or date of last follow-up, assessed up to 5 years
  To assess progression-free survival (PFS) of children with high-grade gliomas treated with a lorlatinib-containing regimen at 1, 3 and 5 years and compare it to historical data from BABYPOG and HIT-SKK.
Associations between genomic tumor alterations with radiographic response | From diagnosis through the end of follow-up period.
  Explore longitudinal associations of genomic, transcriptomic, epigenetic, and/or immunologic alterations of tumor at diagnosis, recurrence, or autopsy with radiographic response and advanced neuro-imaging measures.

CONTACTS AND LOCATIONS:
Overall Officials: Hamza Gorsi, MD, Study Chair — Children's Hospital of Michigan; Susan Chi, MD, Study Chair — Dana-Farber Cancer Institute; Maryam Fouladi, MD, Principal Investigator — Nationwide Children's Hospital
Locations (18):
- United States (10):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University Health System, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Perth Children's Hospital, Perth, Western Australia
- Canada (2):
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- Hopp Children's Cancer Center at NCT Heidelberg (KiTZ), Heidelberg, Baden-Wurttemberg, Germany
- Princess Máxima Center, Utrecht, Netherlands
- Starship Children's Hospital, Auckland, Grafton, New Zealand

IPD SHARING:
Plan to Share IPD: No